CLINICAL TRIAL: NCT06696157
Title: Peer Recovery Support Services (PRSS) for Individuals in Recovery Residences on MOUD (NOTE: EXPANDED SCOPE VERSION OF PROTOCOL)
Brief Title: EXPANDED SCOPE for Parent Grant Entitled, "Peer Recovery Support Services for Individuals in Recovery Residences on MOUD"
Acronym: PRSS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Potomac Health Foundations (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R34DA057627-01-EXPANDED-SCOPE; 1R34DA057627-01 (NIH)
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Opioid Use Disorder
Keywords: Peer Support Specialist; Opioid Use Disorder; Peer Recovery Support Services; Medications for Opioid Use Disorder; MOUD; Substance Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single-arm of an uncontrolled trial of the PRSS intervention for MOUD initiation (Experimental)
  Interventions: Behavioral: PRSS intervention for MOUD initiation

INTERVENTIONS:
Behavioral: PRSS intervention for MOUD initiation — All participants of this expanded scope pilot study will be in a single-arm of an uncontrolled trial of PRSS intervention for MOUD initiation for a total of 8 weeks, starting in inpatient substance abuse treatment. This is distinguished from the R34 parent grant which targets MOUD retention and adherence rather than MOUD initiation.

SUMMARY:
The United States is experiencing an unprecedented opioid epidemic. Medications for opioid use disorder (MOUD), such as methadone, buprenorphine, and extended-release naltrexone, are the recommended standard of care. There are, however, many barriers to MOUD initiation so that only a minority of individuals who could benefit from MOUD treatment ever receive it. Even among individuals presenting to a residential level of specialty SUD care, only about 20% of individuals with OUD initiate MOUD leaving them at a higher risk of opioid relapse, overdose, and death. Thus, the goal of this expansion of scope pilot study is to address this gap by modifying our currently R34-funded intervention (RFA-DA-22-034; Project # 1R34DA057627-01) that leverages the impact of peer recovery support services (PRSS) to promote MOUD initiation. Although PRSS for MOUD initiation shows promise within emergency department settings, the impact of PRSS for MOUD initiation within residential substance use disorder (SUD) settings is unknown. Residential SUD settings are an ideal opportunity to initiate medications because individuals with OUD typically have access to medically-managed withdrawal and the opportunity to learn about and initiate onto MOUD. This PRSS intervention has already been developed in the R34 parent grant to promote MOUD retention, and in this expanded scope project it will be further adapted and tested with a small pilot sample of individuals (N = 10-20) who are further upstream in the cascade of care (COC). Peers will be embedded within the inpatient program unit where the study will take place. Early into their inpatient stay and before MOUD initiation occurs, peers will introduce themselves to patients and provide motivational enhancements for MOUD initiation and inpatient treatment retention through a variety of strategies. Peer strategies will be based on the existing PRSS intervention in the parent grant and may include exploration of MOUD knowledge and attitudes, discussion of relevant lived experience, MOUD psycho-education, and a collaboratively completed wellness plan. Upon discharge, peers will use other strategies to encourage uptake and retention of MOUD such as assertive outreach and emphasize return to care after treatment dropout and/or relapse. The proposed project will explore the feasibility and acceptability of PRSS on MOUD initiation in residential SUD treatment by pilot testing the PRSS intervention with a sample of 10-20 participants receiving an 8-week course of treatment. During the intervention period, the PRSS approach will be adapted and refined with feedback from peer recovery support coaches who have helped develop and test the parent intervention for MOUD retention. Our primary outcomes are: 1) MOUD initiation (yes/no) upon discharge of the inpatient SUD program, and 2) PRSS feasibility and acceptability as measured by a participant satisfaction survey. If this pilot work is successful, the investigators would further test this MOUD initiation-focused version of the PRSS intervention via a future R01-funded Randomized Controlled Trial.

DETAILED DESCRIPTION:
The United States is experiencing an opioid epidemic marked by significant overdose deaths. Although medications for opioid use disorder (MOUD) are efficacious, the rates of MOUD initiation and retention are alarmingly low, with 11% of patients with an OUD diagnosis initiating MOUD and only 3.5% being retained on treatment for a minimum of 6 months. Also, national initiation rates onto MOUD within inpatient substance use disorder (SUD) programs are 18%, which again demonstrates low uptake of MOUD. Supplementing mediation-based treatment with Peer Recovery Support Services (PRSS) may be an effective strategy to encourage MOUD utilization, yet no such evidence-based interventions to specifically improve MOUD initiation and retention currently exist. To address this problem, the ongoing R34 parent grant-funded study (RFA-DA-22-034; Project # 1R34DA057627-01) is developing a new intervention that leverages PRSS to increase MOUD retention in patients living in recovery residences (RRs) and 3.1 residential programs. The parent grant study, however, does not address the aforementioned lagging initiation rates within inpatient SUD treatment programs.

To address this gap, the investigative team is conducting this small pilot study to expand the scope of our parent grant clinical trial to improve MOUD initiation across the OUD cascade of care COC. The ongoing parent grant study's goal is to enhance retention for individuals who have already initiated MOUD and are now living in 3.1 residential programs or Recovery Residences (RRs), which are both further downstream in the OUD COC. This small pilot study will expand the scope of the existing parent project by also utilizing PRSS during inpatient SUD treatment, which is more upstream in the COC.

The rationale for this expansion of scope pilot study is that by recruiting participants who are more stable and further downstream in the OUD COC, the current parent project intervention under investigation misses an opportunity to increase MOUD initiation. Preliminary data gathered from our electronic health record at our institution, Maryland Treatment Centers, showed that only 46% of our inpatients diagnosed with OUD initiate MOUD before leaving inpatient SUD treatment, despite the fact that we recommend MOUD as the first-line standard of care. Furthermore, patients with OUD, which included both premature dropouts and successful program completers, left treatment after an average of two weeks (i.e., 14.89 days). Early dropout limits a patient's opportunities to initiate MOUD and/or become stably retained on MOUD. Thus, investigators will expand the scope of the R34 project to include adapting the existing PRSS intervention for MOUD initiation and obtain pilot data on feasibility in (N = 35) patients enrolled in SUD inpatient treatment. We will accomplish this goal by piloting the PRSS intervention for MOUD initiation during the time that remains for the existing R34 award. All participants will receive the PRSS intervention for a total of 8 weeks.

On important goal of this expanded scope pilot is to explore the feasibility of using PRSS with SUD inpatients. Parent grant Phase 1 qualitative interviews were conducted with stakeholders (N = 16) that included peers (50% of total sample), patients on MOUD (25% of sample), and other professionals working with patients on MOUD (25% of sample) to assess these stakeholders' opinions of the parent grant version of PRSS. Overall, stakeholders found PRSS to be useful and consistent with the tools peers use to help patients adhere to MOUD. The parent grant's rate of recruitment and randomization meets our expected study target goals per month, and demonstrates that the PRSS intervention is feasible with respect to our ability to recruit effectively at Mountain Manor Treatment Center (MMTC), which is under the umbrella of Maryland Treatment Centers and is the study location for this expansion of scope pilot study. Unlike the parent grant that only enrolls patients who are already inducted onto MOUD, this expansion of scope proposal will only recruit people who are in SUD inpatient care and who are not currently on MOUD in an effort to get them to initiate MOUD. In summary, the expanded scope aim is as follows.

Specific Aim: Investigators will pilot an adapted version of the PRSS parent grant intervention that focuses on improving MOUD initiation in a small uncontrolled pilot sample (N = 35) of participants who are being treated further upstream in the OUD COC within an inpatient SUD treatment setting. Hypothesis: Investigators hypothesize that peers and participants will find the modified PRSS intervention to be both acceptable and feasible and that MOUD initiation rates will compare favorably to historical data from our electronic health records.

Impact: The research in this expansion of scope pilot study will contribute to NIDA's overarching mission to ameliorate the ongoing opioid epidemic which continues to be a serious problem in the United States. If successful, this pilot work would be an initial step toward developing an intervention that would help opioid users to initiate MOUD, which is the underutilized standard of care for OUD treatment. This research has great potential to directly reduce the impact of the current opioid epidemic, which is a major public health crisis that continues to plague the USA.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+ (inclusive)
* Meets diagnostic criteria for OUD
* Currently seeking inpatient treatment at Maryland Treatment Centers program
* English speaking
* Willing and able to provide informed consent
* Able to obtain MOUD through insurance.

Exclusion Criteria:

* Having been prescribed and taken a maintenance dose of sublingual buprenorphine or methadone within 14 days of entering the current inpatient treatment episode
* received a dose of XR-buprenorphine or XR-naltrexone within 45 days of entering the current inpatient treatment episode.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-09-29 (Estimated)

PRIMARY OUTCOMES:
MOUD initiation at inpatient substance abuse treatment discharge | 8 weeks
  MOUD initiation status at inpatient substance abuse treatment discharge. Did the participant initiate by the date of discharge? (Yes / No)

SECONDARY OUTCOMES:
MOUD Initiation after inpatient substance use disorder treatment discharge | 8 weeks
  MOUD initiation status at inpatient substance abuse treatment discharge. Did the participant initiate MOUD at any time during the 8 weeks course of the intervention? (Yes / No)
MOUD Retention | 8 weeks
  Among MOUD initiators during inpatient substance abuse treatment, was the participant retained on MOUD at the end of 8 week intervention period? (Yes / No)
Length of inpatient substance abuse treatment stay | 8 weeks
  Number of days retained in inpatient substance abuse treatment care

CONTACTS AND LOCATIONS:
Locations (1):
- Maryland Treatment Centers, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No